CLINICAL TRIAL: NCT02988687
Title: Metabolic and Quality of Life Effects of Growth Hormone Treatment in Patients With Traumatic Brain Injury and AGHD
Brief Title: Metabolic and QOL Effects of GH Treatment in Patients With TBI and AGHD
Status: Completed | Type: Observational
Sponsor: Garcia, Jose M., MD, PhD (Individual)
Responsible Party: Sponsor
Other Study IDs: 00930
Record Dates: First submitted 2016-11-17; First posted 2016-12-09 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2022-08

CONDITIONS: Adult-Onset Growth Hormone Deficiency
Keywords: fatigue; quality of life; depression; cognitive function; growth hormone; traumatic brain injury
MeSH Terms: conditions — Fatigue; Depression; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This PILOT, NON-INTERVENTIONAL STUDY will follow patients about to start rhGH for a period of six months and collect valuable pilot data to evaluate feasibility of a larger study and treatment tolerability and compliance. The effect of rhGH on cognitive function, depression, fatigue, sleep quality, and QOL will also be collected. This exploratory study will also provide important information about recruitment and AGHD screening procedures in military settings.

DETAILED DESCRIPTION:
Growth hormone replacement has consistently shown improvements in body composition, exercise capacity, endothelial function, inflammatory biomarkers, bone mineral density, lipoprotein metabolism, and self-reported quality of Life (QOL) in patients suffering from adult growth hormone deficiency (AGHD). One of the causes for AGHD is traumatic brain injury (TBI), a condition that affects approximately 20% of Veterans from Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND). Because OIF/OEF/OND Veterans are a new population, there is a paucity of data regarding the effects of rhGH in these patients. The investigators propose to perform a pilot observational study of Veterans with confirmed adult growth hormone deficiency (AGHD) due to TBI who have been prescribed recombinant human growth hormone (rhGH) replacement in order to determine changes in metabolic parameters and QOL induced by rhGH.

Our hypothesis is that GH replacement will improve QOL and metabolic parameters (glucose, insulin resistance, lipids, inflammatory markers, and body composition) in patients with confirmed AGHD due to TBI.The primary aim for this proposal is to determine the effects of rhGH treatment given daily for 6 months to Veterans with TBI and AGHD on QoL measured by the Quality of Life Assessment for GHD in Adults questionnaire (QoL-AGHDA, primary outcome). Secondary specific aims for this proposal are to gather high quality pilot data of the effects of 6 months of rhGH replacement in Veterans with TBI and AGHD.

ELIGIBILITY:
Inclusion Criteria:

1. OEF/OIF/OND deployment confirmed by available records
2. history of combat exposure during deployment as determined by a score greater than 1 on the Combat Experiences sub-scale of the Deployment Risk and Resilience Inventory-2 (DRRI-2)
3. age >18 years
4. a history of TBI defined according to the DoD/VA guidelines and characterized by the Ohio State TBI Inventory
5. history of AGH deficiency diagnosed by: a) a GH stimulatory test; or b) low plasma IGF-1 level and 3 pituitary hormone deficiencies
6. have been prescribed rhGH replacement by a clinical provider
7. If the Veteran is receiving psychotropic medications he should be on stable doses for at least 4 weeks before their enrollment in the study.

Exclusion Criteria:

1. Other untreated pituitary deficiencies [patients with other hormone deficiencies will have to be on stable replacement for at least three months before including them on the study; two months of stable replacement is required for hydrocortisone therapy for adrenal insufficiency]
2. tumors, or other causes of AGHD (e.g. childhood onset GHD, pituitary surgery, tumors, radiation)
3. history of neurologic or psychiatric disorder such as stroke, spinal cord injury, bipolar disorder, or schizophrenia that has a significant impact in the Veteran's functional status and QoL
4. contraindication to rhGH therapy (e.g. hypersensitivity to rhGH or any of the components of the supplied product, including metacresol, glycerin, or benzyl alcohol)
5. acute medical illness, active infection, neoplastic disease or decompensated chronic medical illness such as diabetes mellitus (A1c >9%), congestive heart failure or chronic obstructive pulmonary disease
6. evidence of alcohol dependence, alcohol abuse or drug use disorder during the three months previous to enrollment in the study
7. evidence of inadequate levels of effort in performing neuropsychological tests as suggested by scoring less than 41 on Trial I of the Test of Memory and Malingering (TOMM)
8. due to the decreased specificity of the AGHD diagnostic tests in this setting and weight/size limitations of the DEXA scanner, we will exclude morbid obese subjects defined as having a BMI greater than 35 or body weight > 350 lbs
9. use of rhGH in the previous 6 months
10. active or recent (6 months) history of coronary artery or cerebrovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans being prescribed rhGH replacement for Adult Onset Growth Hormone Deficiency due to Traumatic Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-11; Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
AGHDA change | baseline to 3 months
  Quality of Life Assessment for GHD in Adults questionnaire
AGHDA change | baseline to 6 months
  Quality of Life Assessment for GHD in Adults questionnaire

SECONDARY OUTCOMES:
Body composition change | baseline to 6 months
  Lean body mass and fat mass by dual energy x-ray absorptiometry
CVLT change | baseline to 6 months
  Memory performance measured by the California Verbal Learning
DASS-21 change | baseline to 6 months
  Depressive and anxiety symptoms measured by the Depression Anxiety and Stress Scale

OTHER OUTCOMES:
muscle strength change | baseline to 6 months
  1-RM and hand grip strength (both in kg)
Aerobic capacity change | baseline to 6 months
  VO2 max
Muscle function change | baseline to 6 months
  chair stand test
Muscle function change | baseline to 6 months
  stair climb power
Fatigue change | baseline to 6 months
  QOL AGHD subsection
Sleep quality change | baseline to 6 months
  Pittsburgh Sleep Quality Index
Inflammatory marker changes | baseline to 6 months
  systemic cytokine levels
Anabolic marker changes | baseline to 6 months
  systemic IGF-1 and IGFBP3 levels (both ng/mL)
Chronic pain change | baseline to 6 months
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herodes M, Le N, Anderson LJ, Migula D, Miranda G, Paulsen L, Garcia JM. Metabolic and quality of life effects of growth hormone replacement in patients with TBI and AGHD: A pilot study. Growth Horm IGF Res. 2023 Aug;71:101544. doi: 10.1016/j.ghir.2023.101544. Epub 2023 Jun 1. PMID 37295336